CLINICAL TRIAL: NCT03290781
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Study of SHP647 as Maintenance Therapy in Subjects With Moderate to Severe Ulcerative Colitis (FIGARO UC 303)
Brief Title: An Efficacy and Safety Study of Ontamalimab as Maintenance Therapy in Participants With Moderate to Severe Ulcerative Colitis
Acronym: FIGARO UC 303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP647-303; 2017-000573-37 (EudraCT Number)
Record Dates: First submitted 2017-09-06; First posted 2017-09-25 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ontamalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ontamalimab 25 mg (Experimental): Participants will receive 25 milligram (mg) of ontamalimab or placebo and achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) will receive 25 mg of ontamalimab as maintenance treatment subcutaneously using a prefilled syringe once in every 4 weeks (Q4W) up to Week 52.
  Interventions: Drug: Ontamalimab
- Ontamalimab 75 mg (Experimental): Participants will receive 75 mg of ontamalimab or placebo and achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) will receive 75 mg of ontamalimab as maintenance treatment subcutaneously using a prefilled syringe Q4W up to Week 52.
  Interventions: Drug: Ontamalimab
- Placebo (Placebo Comparator): Participants will receive 25 mg or 75 mg ontamalimab or placebo matched to ontamalimab in the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) will receive placebo matched to ontamalimab as maintenance treatment subcutaneously using a prefilled syringe Q4W up to Week 52.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ontamalimab — Participants will receive 1 milliliter (mL) of ontamalimab sterile aqueous buffered solution at an appropriate oncentration to provide an intended dose of drug (25 or 75 mg).
  Other Names: PF-00547659; SHP647
  Arms: Ontamalimab 25 mg; Ontamalimab 75 mg
Other: Placebo — Participants will receive 1 mL of sterile aqueous buffered solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ontamalimab as maintenance therapy treatment of remission, based on composite score of patient-reported symptoms and centrally read endoscopy, in participants with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or their parent or legally authorized representative must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Participants must be able to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent and/or assent, as applicable, to participate in the study.
* Participants must have completed the 12-week induction treatment period (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]).
* Participants must have achieved clinical response in induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]). Clinical response is defined as:

  i) A decrease from the induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) baseline in the composite score of patient reported symptoms using daily e-diary and centrally read endoscopy of at least 2 points and at least 30 percent (%), with an accompanying decrease in the sub score for rectal bleeding greater than or equal to (>=) 1 point or a sub score for rectal bleeding less than or equal to (<=) 1 OR ii) A decrease from the induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) baseline in total Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the rectal bleeding sub score of at least 1 point or an absolute rectal bleeding sub score of 0 or 1.

For eligibility assessment, clinical response will be determined based on the centrally read endoscopy performed during screening and at Week 12 of induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]).

- Participants receiving any treatment(s) for ulcerative colitis (UC) are eligible provided they have been, and are anticipated to be, on a stable dose for the designated period of time.

Exclusion Criteria:

* Participants who had major protocol deviation(s) (as determined by the sponsor) in induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]).
* Participants who permanently discontinued investigational product because of an adverse event (AE), regardless of relatedness to investigational product, in induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]).
* Participants who are likely to require surgery for UC during the study period.
* Participants are females who became pregnant during induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]), females who are planning to become pregnant during the study period, or males or females of childbearing potential not agreeing to continue using appropriate contraception methods (that is [i.e,] highly effective methods for female and medically appropriate methods for male study participants) through the conclusion of study participation.
* Participants who do not agree to postpone donation of any organ or tissue, including male participants who are planning to bank or donate sperm and female participants who are planning to harvest or donate eggs, for the duration of the study and through 16 weeks after last dose of investigational product.
* Participants who, in the opinion of the investigator or the sponsor, will be uncooperative or unable to comply with study procedures.
* Participants who have a newly diagnosed malignancy or recurrence of malignancy (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
* Participants who have developed any major illness/condition or evidence of an unstable clinical condition (example [eg], renal, hepatic, hematologic, gastrointestinal (except disease under study), endocrine, cardiovascular, pulmonary, immunologic [eg, Felty's syndrome], or local active infection/infectious illness) that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study.
* Participants with any other severe acute or chronic medical or psychiatric condition or laboratory or electrocardiogram (ECG) abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participants with known exposure to Mycobacterium tuberculosis (TB) since testing at screening in induction study (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) and who are without a generally accepted course of treatment.
* Participants who are investigational site staff members or relatives of those site staff members or participants who are sponsor employees directly involved in the conduct of the study.
* Participants who are participating in or plan to participate in other investigational studies (other than induction study SHP647- 301 [NCT03259334] and SHP647-302 [NCT03259308]) during study SHP647-303 [NCT03290781].

Ages: 16 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (399):
- United States (93):
  - Arizona Digestive Health Mesa - East, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - Clinedge - PPDS, Phoenix, Arizona
  - Atria Clinical Research - Clinedge - PPDS, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - United Medical Doctors, Encinitas, California
  - University of California San Diego, La Jolla, California
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - VA Long Beach Healthcare System - NAVREF - PPDS, Long Beach, California
  - Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - Alliance Clinical Research-(Vestavia Hills), Poway, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California San Francisco, San Francisco, California
  - Care Access Research, San Pablo, San Pablo, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Asthma and Allergy Associates PC - CRN - PPDS, Colorado Springs, Colorado
  - Renaissance Research Medical Group, INC, Cape Coral, Florida
  - Gastro Florida, Clearwater, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Alliance Medical Research LLC, Coral Springs, Florida
  - ENCORE Borland-Groover Clinical Research - ERN - PPDS, Jacksonville, Florida
  - SIH Research, Kissimmee, Florida
  - Hi Tech and Global Research, LLc, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Pharma Research International Inc, Naples, Florida
  - Omega Research Consultants LLC - Clinedge - PPDS, Orlando, Florida
  - Accel Research Sites - St. Petersburg - ERN - PPDS, Pinellas Park, Florida
  - BRCR Medical Center, Inc, Plantation, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - DBC Research, Tamarac, Florida
  - Bayside Clinical Research - New Port Richey, Tampa, Florida
  - Atlanta Gastroenterology Specialists, PC, Atlanta, Georgia
  - Infinite Clinical Trials, Atlanta, Georgia
  - Gastrointestinal Diseases, Inc Research - IACT- HyperCore - PPDS, Columbus, Georgia
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Loretto Hospital, Chicago, Illinois
  - IL Gastroenterology Group, Gurnee, Illinois
  - Edward Hines Jr VA Hospital - NAVREF - PPDS, Hines, Illinois
  - Dupage Medical Group, Oakbrook Terrace, Illinois
  - Medisphere Medical Research Center LLC, Evansville, Indiana
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - CroNOLA, LLC., Houma, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Commonwealth Clinical Studies LLC, Brockton, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Mayo Clinic Health System - PPDS, Duluth, Minnesota
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - St Louis Center For Clinical Research, St Louis, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Encompass Care, North Las Vegas, Nevada
  - New York Total Medical Care PC, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - Weill Cornell Medical College, New York, New York
  - Southtowns Gastroenterology, PLLC, Orchard Park, New York
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Consultants For Clinical Research Inc, Fairfield, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Ohio Clinical Research Partners LLC, Mentor, Ohio
  - Veteran's Research and Education Foundation - NAVREF - PPDS, Oklahoma City, Oklahoma
  - Veterans Research Foundation of Pittsburgh - NAVREF - PPDS, Pittsburgh, Pennsylvania
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology-Union City, Union City, Tennessee
  - Inquest Clinical Research/Coastal Gastroenterology Associates, PA - TDDC - PPDS, Baytown, Texas
  - Northside Gastroenterology, Cypress, Texas
  - Digestive Health Associates of Texas, P.A.dba DHAT Research Institute, Garland, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Aztec Medical Research, Houston, Texas
  - BI Research Center, Houston, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - HP Clinical Research, Bountiful, Utah
  - Mid Atlantic Health Specialists, Galax, Virginia
  - Winchester Gastroenterology Associates, Winchester, Virginia
  - CHI Franciscan Digestive Care Associates, Tacoma, Washington
  - Exemplar Research, Inc. - Elkins, Elkins, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Argentina (3):
  - Fundación Favaloro, Buenos Aires
  - Hospital Privado Centro Médico de Córdoba, Córdoba
  - Sanatorio 9 de Julio SA, San Miguel de Tucumán
- Australia (7):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Box Hill, Victoria
  - St Vincents Hospital Melbourne - PPDS, Melbourne, Victoria
- Austria (7):
  - A.ö. Krankenhaus der Barmherzigen Brüder, Sankt Veit an der Glan, Carinthia
  - Universitätsklinikum St. Pölten, Sankt Pölten, Saint Pölten
  - LKH-Universitätsklinikum Klinikum Graz, Graz, Styria
  - Klinikum Klagenfurt Am Woerthersee, Klagenfurt
  - Salzburger Landeskliniken, Salzburg
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (4):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Gasthuisberg, Leuven, Vlaams Brabant
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - CHU Mouscron, Mouscron
- Clinical Center Banja Luka, Banja Luka, Bosnia and Herzegovina
- Bulgaria (13):
  - University Multiprofile Hospital for Active Treatment Sveta Anna, Sofia, Sofia-Grad
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski EAD, Pleven
  - Multiprofile Hospital for Active Treatment Eurohospital, Plovdiv
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases Dr.D.Gramatikov- Ruse- PPDS, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Convex EOOD, Sofia
  - Diagnostic Consultative Centre Mladost - M OOD, Varna
- Canada (2):
  - Percuro Clinical Research LTD, Victoria, British Columbia
  - Toronto Digestive Disease Associates Inc, Toronto, Ontario
- Colombia (3):
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Servimed S.A.S, Bucaramanga, Santander Department
  - IPS Centro Médico Julián Coronel S.A.S. - PPDS, Cali
- Croatia (8):
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - Opca Bolnica Karlovac, Karlovac, Karlovacka Županija
  - Opca bolnica Bjelovar, Bjelovar
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital Centre Split, Split
  - General Hospital Virovitica, Virovitica
  - General County Hospital Vukovar and Croatian Veterans Hospital, Vukovar
  - General Hospital Zadar, Zadar
- Czechia (6):
  - Hepato-Gastroenterologie HK, s. r. o., Hradec Králové, Královéhradecký kraj
  - PreventaMed s.r.o., Olomouc, Olomoucký kraj
  - Institut Klinicke A Experimentalni Mediciny, Prague
  - ISCARE I.V.F. a.s., Prague
  - Nemocnice Pardubickeho kraje, a.s. Orlickoustecka nemocnice, Ústi Nad Orlici
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Estonia (3):
  - East Viru Central Hospital, Kohta-Järve
  - OÜ LV Venter, Pärnu
  - West Tallinn Central Hospital, Tallinn
- Germany (12):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Gastro Campus Research GbR, Münster, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitatsklinikum Jena, Jena, Thuringia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Gastroenterologische Facharztpraxis am Mexikoplatz, Berlin-Zehlendorf
  - Sana Klinikum Biberach, Biberach an der Riss
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Westklinikum Hamburg Ggmbh, Hamburg
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, Munich
- Greece (4):
  - Ippokrateio General Hospital of Athens, Athens, Attica
  - University General Hospital of Patras, Pátrai
  - Theageneio Anticancer Oncology Hospital of Thessaloniki, Thessaloniki
  - Euromedica - PPDS, Thessaloniki
- Hungary (12):
  - Bekes Megyei Kozponti Korhaz, Békéscsaba
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - ENDOMEDIX Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz, Gyula
  - Mohacsi Korhaz, Mohács
  - Tolna Megyei Balassa János Kórház, Szekszárd
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Jávorszky Ödön Kórház, Vác
  - Csolnoky Ferenc Korhaz, Veszprém
- St Vincent's University Hospital, Dublin, Ireland
- Israel (6):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem
  - Galilee Medical Center, Nahariya
  - Nazareth EMMS Hospital, Nazareth
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
  - Baruch Padeh Poriya Medical Center, Tiberias
- Italy (15):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera Mater Domini Di Catanzaro, Catanzaro, Calabria
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
  - Azienda Ospedale Università Padova - Dipartimento Salute della Donna e del Bambino, Padua, Veneto
  - A.O.U. Maggiore della Carità, Novara
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - La Sapienza-Università di Roma-Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Japan (34):
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Medical Corporation Aoyama Clinic, Kobe, Hyôgo
  - Hyogo College of Medicine, Nishinomiya-shi, Hyôgo
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Nihonbashi Egawa Clinic, Chuo-Ku, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Ome Municipal General Hospital, Ōme, Tokyo
  - Tokatsu Tsujinaka Hospital, Abiko
  - Kunimoto Hospital, Asahikawa
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hakodate Koseiin Hakodate Goryoukaku Hospital, Hakodate
  - Yuai Memorial Hospital, Koga
  - Kawabe Clinic, Koganei
  - Hidaka Coloproctology Clinic, Kurume-shi
  - Aizawa Hospital, Matsumoto-shi
  - Aichi Medical University Hospital, Nagakute
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Onomichi General Hospital, Onomichi
  - Chiinkai Dojima General & Gastroenterology Clinic, Osaka
  - Kinshukai Infusion Clinic, Osaka
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Shiga University of Medical Science Hospital, Ōtsu
  - Bellland General Hospital, Sakai
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Sapporo Tokushukai Hospital, Sapporo
  - Tohoku Rosai Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga-gun
  - Medical Corporation Shoyu-kai Fujita Gastroenterology Hospital, Takatsuki
  - Koukokukai Ebisu Clinic, Tokyo
  - Shinbeppu Hospital, Beppu, Ôita
  - Yodogawa Christian Hospital, Osaka, Ôsaka
- Lebanon (2):
  - Rafik Hariri University Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - Vilnius City Clinical Hospital, Vilnius
- Mexico (10):
  - Clinica de Higado y Gastroenterologia Integral, S.C., Cuernavaca, Morelos
  - JM Research S.C, Cuernavaca, Morelos
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Centro de Investigación Médica Aguascalientes, Aguascalientes
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli
  - Centro de Investigacion Clinica Acelerada, S.C., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Accelerium, S. de R.L. de C.V., Monterrey
  - Clinical Research Institute, Tlalnepantla
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan
- Netherlands (5):
  - ETZ-Elisabeth, Tilburg, North Brabant
  - NWZ, location Alkmaar, Alkmaar, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - VU Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum Amsterdam, Amsterdam
- New Zealand (4):
  - Auckland City Hospital, Grafton, Auckland
  - Dunedin Hospital, Dunedin, South Island
  - Wellington Hospital, Newtown, Wellington Region
  - Waikato Hospital, Hamilton
- Poland (36):
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp.j.Specjalistyczne Centrum Gastrologii i Endoskopii Specj, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o., Włocławek, Kuyavian-Pomeranian Voivodeship
  - Krakowskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Lexmedica, Wroclaw, Lower Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lódz, Lódzkie
  - Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Centralny Szpital Weteranow, Lódz, Lódzkie
  - Instytut Centrum Zdrowia Matki Polki, Lódz, Lódzkie
  - BioVirtus Centrum Medyczne, Józefów, Masovian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej VIVAMED, Warsaw, Masovian Voivodeship
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Szpital Zakonu Bonifratrow pw. Aniolow Strozow w Katowicach, Katowice, Silesian Voivodeship
  - Twoja Przychodnia - Szczecińskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Czestochowa - PRATIA - PPDS, Częstochowa
  - Centrum Medyczne Gdynia - PRATIA - PPDS, Gdynia
  - NZOZ All Medicus, Katowice
  - Centrum Medyczne A-Z Clinic Mateusz Sidor, Piotr Puc-Lekarze Spolka Partnerska, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Med Gastr Sp.z.o.o Sp.k, Lodz
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Centrum Innowacyjnych Terapii, Piaseczno
  - Clinical Research Center Spółka z Ograniczoną Odpowiedzialnością, Medic-R Spółka Komandytowa, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Bandurskiego 98/U12, Szczecin
  - Sonomed Sp. z o.o., Szczecin
  - H-T. Centrum Medyczne Endoterapia, Tychy
  - Centrum Zdrowia MDM, Warsaw
  - Centrum Medyczne Warszawa - PRATIA - PPDS, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość
  - Szpital Specjalistyczny sw Lukasza - Oddzial Gastroenterologii, Gmina Końskie, Świętokrzyskie Voivodeship
- Portugal (5):
  - Hospital da Luz, Lisbon, Lisbon District
  - Hospital de Braga, Braga
  - Centro Hospitalar do Algarve - Hospital de Portimao, Faro
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Hospital de São Bernardo, Setúbal
- Romania (11):
  - Cluj-Napoca Emergency Clinical County Hospital, Cluj-Napoca, Cluj
  - Dr.Carol Davila Emergency University Central Military Hospital, Bucharest
  - Sana Monitoring SRL, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Centrul Medical Hifu Terramed Conformal S.R.L., Bucharest
  - Affidea Romania SRL, Constanța
  - Gastromedica SRL, Iași
  - Dr. Tirnaveanu Amelita Private Practice, Oradea
  - Dr. Goldis Gastroenterology Center SRL, Timișoara
- Russia (17):
  - Kazan State Medical University, Kazan'
  - Moscow Clinical Scientific Center, Moscow
  - Moscow Regional Research Clinical Institute Na Mfvladimirskiy, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Research Institute of Physiology and Basic Medicine, Novosibirsk
  - Rostov State Medical University, Rostov-on-Don
  - St. Elizabeth Municipal Clinical Hospital, Saint Petersburg
  - First St. Petersburg State Medical University n.a. I.P Pavlov, Saint Petersburg
  - Union Clinic, LLC, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Medical University Reaviz, Samara
  - Private Healthcare Institution Clinical Hospital RZD-Medicina of Samara city, Samara
  - Medical Company Hepatolog, LLC, Samara
  - SHI Regional Clinical Hospital, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - Stavropol State Medical University, Stavropol
  - Regional Consulting and Diagnostics Centre, Tyumen
- Serbia (4):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - University Clinical Center Nis, Niš
  - General Hospital Vrsac, Vršac
  - University Clinical Center Kragujevac, Kragujevac, Šumadijski Okrug
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava
  - KM Management, spol. s r.o., Nitra
  - Gastro LM, s.r.o., Prešov
- South Africa (3):
  - CLINRESCO, ARWYP Medical Suites, Johannesburg, Gauteng
  - Dr. J Breedt, Pretoria, Gauteng
  - Dr JP Wright, Claremont, Western Cape
- South Korea (16):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang'yeogsi
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gang'weondo
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeonggido
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center PPDS, Seoul
  - Inje University Seoul Paik Hospital, Seoul
- Spain (10):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Centro Medico Teknon - Grupo Quironsalud, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universität Zürich, Zurich, Zürich (de), Switzerland
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Mersin University Medical Faculty, Mersin
- Ukraine (25):
  - Regional Municipal Non-profit Enterprise "Chernivtsi Regional Clinical Hospital", Chernivtsi, Chernivtsi Oblast
  - Municipal Nonprofit Enterprise CCH #2 n.a. prof. O.O. Shalimov of Kharkiv City Council, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv, Kyïv
  - Communal Nonprofit Enterprise Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VRC, Vinnytsia, Vinnytsia Oblast
  - Municipal Non-profit Enterprise City Emergency Care Hospital of Zaporizhzhia Regional Council, Zaporizhzhia, Zaporizhzhia Oblast
  - ME Dnipropetrovsk Regional Clinical Hospital n.a. I.I Mechnykov Dnipropetrovsk Regional Council, Dnipro
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipro
  - Clinic of SI National Institute of Therapy n.a. L.T. Mala of NAMS of Ukraine, Kharkiv
  - Communal Non-Commercial Enterprize of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - MNPE of Kharkiv Regional Council Regional Clinical Specialized Dispensary of Radiation Protection, Kharkiv
  - Municipal Non-profit Enterprise Kherson City Clinical Hospital named after Ye.Ye. Karabelesh, Kherson
  - Municipal Enterprise Kryvyi Rih City Clinical Hospital #2 of Kryvyi Rih City Council, Kryvyi Rih
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv
  - Kyiv City Clinical Hospital #18, Kyiv
  - Treatment and Diagnostic Center "Healthy and Happy" of LLC "Healthy and Happy", Kyiv
  - Municipal Institution of KRC Kyiv Regional Hospital #2, Kyiv
  - Lviv Railway Clinical Hospital of branch Health Center of Joint Stock Co. Ukrainian Railway, Lviv
  - Municipal Nonprofit Enterprise Lviv Clinical Emergency Care Hospital, Lviv
  - Municipal Non-profit Enterprise Odessa Regional Clinical Hospital of Odessa Regional Council, Odesa
  - MNPE Central City Clinical Hospital of Uzhhorod City Council, Uzhhorod
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
  - Communal Nonprofit Enterprise Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VRC, Vinnytsia
  - Communal Non-Commercial Enterprise Vinnytsia City Clinical Hospital 1, Vinnytsia
  - MNPE City Hospital No. 6 of Zaporizhzhia City Council, Zaporizhzhia
- United Kingdom (8):
  - Aberdeen Royal Infirmary - PPDS, Aberdeen, Aberdeen City
  - Fairfield General Hospital - PPDS, Lancashire, Bury
  - Whipps Cross University Hospital, London, London, City of
  - North Tyneside General Hospital, North Shields, Northumberland
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - Western General Hospital Edinburgh - PPDS, Edinburh
  - Royal Gwent Hospital - PPDS, Newport
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Vermeire S, Danese S, Sandborn WJ, Schreiber S, Hanauer S, D'Haens G, Nagy P, Thakur M, Bliss C, Cataldi F, Goetsch M, Gorelick KJ, Reinisch W. Efficacy and Safety of the Anti-mucosal Addressin Cell Adhesion Molecule-1 Antibody Ontamalimab in Patients with Moderate-to-Severe Ulcerative Colitis or Crohn's Disease. J Crohns Colitis. 2024 May 31;18(5):708-719. doi: 10.1093/ecco-jcc/jjad199. PMID 38096402
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdf4db2bf003ab47502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 400 sites from 4 April 2018 (first participant first visit) to 1 July 2021 (last participant last visit). A total of 366 participants were enrolled, randomized and received study treatment.
Pre-assignment Details: Participant with moderate to severe Ulcerative Colitis (UC) who achieved a clinical response and completed their treatment period in the induction studies (either SHP647-301 [NCT03259334] or SHP647-302 [NCT03259308]) were randomized into this study as ontamalimab and placebo responders to receive placebo or ONTA 25 milligrams (mg) or 75 mg.
Groups:
- ONTA 25mg/ Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in every 4 weeks (Q4W) up to Week 52.
- ONTA 25mg/ONTA 25mg: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive 25 mg of ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- ONTA 75mg/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 75 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- ONTA 75mg/ONTA 75mg: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 75 mg of ontamalimab were randomized to receive 75 mg of ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- Placebo/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with placebo were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- Placebo/ONTA 25mg: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with placebo were randomized to receive 25 mg of ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- Placebo/ONTA 75mg: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with placebo were randomized to receive 75 mg of ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
Period: Overall Study
Arm/Group | ONTA 25mg/ Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg | Placebo/Placebo | Placebo/ONTA 25mg | Placebo/ONTA 75mg
Started | 73 | 71 | 86 | 82 | 11 | 22 | 21
Completed | 24 | 53 | 30 | 59 | 6 | 19 | 17
Not Completed | 49 | 18 | 56 | 23 | 5 | 3 | 4
Not completed — Adverse Event | 5 | 7 | 4 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 9 | 10 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 1 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Disease Relapse | 32 | 5 | 38 | 7 | 3 | 1 | 4
Not completed — Other | 3 | 0 | 2 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who had received at least 1 dose of Investigational Product (IP) in this study, regardless of treatment received during the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]).
Groups:
- ONTA 25mg/ Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- ONTA 75mg/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 75 mg of ontamalimab were randomized to receive placebo matched to ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- Total: Total of all reporting groups
Arm/Group | ONTA 25mg/ Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg | Placebo/Placebo | Placebo/ONTA 25mg | Placebo/ONTA 75mg | Total
Number analyzed (Participants) | 73 | 71 | 86 | 82 | 11 | 22 | 21 | 366
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (15.40) | 41.2 (13.17) | 42.0 (13.81) | 42.3 (14.21) | 44.7 (14.16) | 40.9 (9.42) | 39.9 (12.10) | 42.1 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 35 | 35 | 5 | 9 | 10 | 150
  Male | 46 | 42 | 51 | 47 | 6 | 13 | 11 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 4 | 7 | 0 | 3 | 1 | 27
  Not Hispanic or Latino | 67 | 64 | 82 | 74 | 11 | 19 | 20 | 337
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 4
  Asian | 5 | 4 | 5 | 8 | 1 | 2 | 3 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 1 | 2 | 2 | 0 | 0 | 1 | 9
  White | 58 | 62 | 77 | 69 | 10 | 19 | 17 | 312
  More than one race | 4 | 2 | 0 | 0 | 0 | 1 | 0 | 7
  Unknown or Not Reported | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Remission Based on Composite Score at Week 52
Description: Remission: a composite score of participant reported symptoms using daily e-diary and centrally read endoscopy as follows: stool frequency sub-score 0 or 1 with at least a 1-point change from induction study baseline; and rectal bleeding sub-score of 0; and endoscopic sub-score 0 or 1 (modified, excludes friability). The composite score was a recommended measure consisted of Mayo score without the Physician global assessment (PGA) sub-score and ranges from 0-9 points. The Mayo score was a measure of UC disease activity ranged from 0-12 points and consisted of 4 sub-scores, each graded from 0-3 with higher scores indicating more severe disease. Sub-scores were rectal bleeding (range: 0-3, where 0= no blood & 3=blood alone passes), stool frequency (range: 0-3, where 0= normal number of stools and 3=at least 5 stools more than normal), PGA sub-score (range: 0-3- higher score= severe disease), and an endoscopic sub-score (range: 0-3, where 0= normal/inactive disease; 3= severe disease).
Time Frame: At Week 52
Population: The ontamalimab responder full analysis set (FAS) consisted of all participants in the randomized set who received at least 1 dose of IP in this study and who were previously treated with ontamalimab in the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]). As Pre-specified in protocol all efficacy analyses data were collected and analyzed based on ontamalimab responder (i.e ONTA 25mg/ Placebo, ONTA 25mg/ONTA 25mg, ONTA 75mg/Placebo and ONTA 75mg/ONTA 75mg arms only).
Measure: Count of Participants; unit: Participants
Groups:
- ONTA 25 mg/ Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- ONTA 25 mg/ONTA 25 mg: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive 25 mg of ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- ONTA 75 mg/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 75 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
- ONTA 75 mg/ONTA 75 mg: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 75 mg of ontamalimab were randomized to receive 75 mg of ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
Arm/Group | ONTA 25 mg/ Placebo | ONTA 25 mg/ONTA 25 mg | ONTA 75 mg/Placebo | ONTA 75 mg/ONTA 75 mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 6 | 38 | 11 | 33
Statistical Analysis 1: Comparison: ONTA 25 mg/ Placebo vs ONTA 25 mg/ONTA 25 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value was based on CMH chi-square test stratified by status of glucocorticoid use at SHP647-303 baseline, prior anti-TNF treatment, and the degree of clinical response in the induction studies (whether remission is achieved or not); Difference in Proportion = 0.451, 95% CI 2-sided [0.296 to 0.572]
Statistical Analysis 2: Comparison: ONTA 75 mg/Placebo vs ONTA 75 mg/ONTA 75 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.278, 95% CI 2-sided [0.142 to 0.401]

2. Secondary Outcome: Number of Participants With Endoscopic Remission at Week 52
Description: Endoscopic remission was defined by centrally read endoscopic sub-score 0 or 1 (modified, excludes friability). The centrally read endoscopic sub-score of mayo score ranged from 0 to 3, where 0=normal or inactive disease; 3=severe disease (spontaneous bleeding, ulceration).
Time Frame: At Week 52
Population: The ontamalimab responder FAS consisted of all participants in the randomized set who received at least 1 dose of IP in this study and who were previously treated with ontamalimab in the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]). As Pre-specified in protocol all the efficacy analyses data were collected and analyzed based on ontamalimab responder FAS only (i.e ONTA 25mg/ Placebo, ONTA 25mg/ONTA 25mg, ONTA 75mg/Placebo and ONTA 75mg/ONTA 75mg).
Measure: Count of Participants; unit: Participants
Groups:
- ONTA 25mg/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 7 | 40 | 13 | 40
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.463, 95% CI 2-sided [0.310 to 0.585]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.339, 95% CI 2-sided [0.197 to 0.463]

3. Secondary Outcome: Number of Participants With Clinical Remission at Week 52
Description: Clinical remission was defined by stool frequency sub-score of 0 or 1 with at least a 1-point change from induction study baseline in stool frequency sub-score, and rectal bleeding sub-score of 0. Rectal bleeding was assessed on a scale from 0-3, where 0: no blood seen, 1: streaks of blood with stool less than half time, 2: obvious blood or streaks of blood with stool most of the time, and 3: blood alone passes. Stool frequency was assessed on a scale from 0-3, where 0: normal number of stools for this participant, 1: 1 to 2 stools more than normal; 2: 3 to 4 stools more than normal, and 3: 5 or more stools more than normal. Higher scores indicated more severe disease.
Time Frame: At Week 52
Population: The ontamalimab responder FAS consisted of all participants in the randomized set who received at least 1 dose of IP in this study and who were previously treated with ontamalimab in the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]). As Pre-specified in protocol all the efficacy analyses data were collected and analyzed based on ontamalimab responder (i.e ONTA 25mg/ Placebo, ONTA 25mg/ONTA 25mg, ONTA 75mg/Placebo and ONTA 75mg/ONTA 75mg arms only).
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 13 | 48 | 19 | 42
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.497, 95% CI 2-sided [0.337 to 0.620]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.294, 95% CI 2-sided [0.148 to 0.425]

4. Secondary Outcome: Number of Participants With Sustained Remission at Week 52
Description: Sustained remission was defined as in remission at Week 52 visit, among participants who were in remission at the time of baseline. Remission was defined as a stool frequency sub-score of 0 or 1 with at least a 1-point change from induction study baseline in stool frequency sub-score and rectal bleeding sub-score of 0 and endoscopic sub-score of 0 or 1 (modified, excludes friability). Sub-scores were rectal bleeding (range: 0-3, where 0= no blood & 3=blood alone passes), stool frequency (range: 0-3, where 0= normal number of stools and 3=at least 5 stools more than normal), and an endoscopic sub-score (range: 0-3, where 0= normal/inactive disease; 3= severe disease).
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 4 | 23 | 7 | 22
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.277, 95% CI 2-sided [0.129 to 0.398]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.191, 95% CI 2-sided [0.067 to 0.305]

5. Secondary Outcome: Number of Participants With Clinical Response Based on Composite Score at Week 52
Description: Clinical response was defined as a decrease from induction study baseline in the composite score of subject reported symptoms using daily e-diary and centrally read endoscopy of at least 2 points and at least 30%, with an accompanying decrease in the sub-score for rectal bleeding >=1 point or a sub-score for rectal bleeding <= 1. Composite score consisted of Mayo score without the PGA sub-score and ranges from 0 to 9 points. Mayo score was a measure of UC disease activity, ranged from 0 -12 points and consisted of 4 sub-scores, each graded from 0 -3, higher scores indicating more severe disease. The rectal bleeding sub-scores ranges from 0-3, where 0= no blood & 3=blood alone passes and centrally read endoscopic sub-score ranges from 0-3, where 0= normal/inactive disease; 3= severe disease.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 15 | 49 | 20 | 47
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.488, 95% CI 2-sided [0.329 to 0.613]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.343, 95% CI 2-sided [0.194 to 0.471]

6. Secondary Outcome: Number of Participants With Mucosal Healing Based on Endoscopic and Histologic Assessment at Week 52
Description: Mucosal healing was defined by centrally read endoscopic sub-score 0 or 1 (modified, excludes friability) and centrally read Geboes score of <=2. The centrally read endoscopic sub-score of mayo score ranges from 0 to 3 with higher scores indicating more severe disease. Geboes score grading system, was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicates more severe disease.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 6 | 37 | 11 | 29
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.431, 95% CI 2-sided [0.280 to 0.554]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.227, 95% CI 2-sided [0.094 to 0.349]

7. Secondary Outcome: Number of Participants With Glucocorticoid-free Clinical Remission at Week 52
Description: Glucocorticoid-free clinical remission was defined as clinical remission in addition to not requiring any treatment with glucocorticoids for at least 4 weeks prior to the Week 52 visit among participants using glucocorticoids at the baseline. Clinical remission was defined as stool frequency sub-score of 0 or 1 with at least a 1-point change from induction study baseline in stool frequency sub-score, and rectal bleeding sub-score of 0, at the Week 52 visit. The stool frequency sub-score ranges from 0-3, where 0= normal number of stools and 3=at least 5 stools more than normal and rectal bleeding sub-score ranges from 0-3, where 0= no blood & 3=blood alone passes).
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- ONTA 25mg/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive placebo matched to ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 1 | 12 | 3 | 12
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.176, 95% CI 2-sided [0.049 to 0.287]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p < 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Proportion = 0.111, 95% CI 2-sided [0.006 to 0.208]

8. Secondary Outcome: Number of Participants With Glucocorticoid-free Remission at Week 52
Description: Glucocorticoid-free remission was defined as remission in addition to not requiring any treatment with glucocorticoids for at least 4 weeks prior to the Week 52 visit, among participants using glucocorticoids at the baseline. Remission was defined as a composite score of participant-reported symptoms using daily e-diary and endoscopy, with stool frequency sub-score of 0 or 1 with at least a 1-point change from induction study baseline, and rectal bleeding sub-score of 0, and endoscopic sub-score of 0 or 1 (modified, excludes friability). The composite score was a recommended measure consisting of the Mayo score without the PGA sub-score and ranges from 0 to 9 points. The stool frequency sub-score, rectal bleeding sub-score and endoscopic sub-score of mayo score ranges from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 0 | 8 | 2 | 10
Statistical Analysis 1: Comparison: ONTA 25mg/Placebo vs ONTA 25mg/ONTA 25mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ONTA 75mg/Placebo vs ONTA 75mg/ONTA 75mg; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel — P-value was based on CMH chi-square test stratified by status of glucocorticoid use at SHP647- 303 baseline, prior anti-TNF treatment, and the degree of clinical response in the induction studies (whether remission is achieved or not)

9. Secondary Outcome: Number of Participants With Remission Based on Total Mayo Score at Week 52
Description: Remission defined as a total mayo score of less than or equal to (<=) 2 with no individual sub-score (stool frequency, rectal bleeding, endoscopy [modified, excludes friability], and physician's global assessment) exceeding 1. The total mayo score ranges from 0 to 12 points and consisted of the following 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: Sub-scores were rectal bleeding (range: 0 to 3, where 0=no blood seen and 3=blood alone passes), stool frequency (range: 0 to 3, where 0=normal number of stools and 3=at least 5 stools more than normal), PGA sub-score (range: 0 to 3-higher score indicating the severe disease), and an endoscopic sub-score (range: 0 to 3, where 0=normal or inactive disease; 3=severe disease [spontaneous bleeding, ulceration].
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 5 | 38 | 10 | 33

10. Secondary Outcome: Number of Participants With Clinical Remission Based on Both Rectal Bleeding and Stool Frequency Sub-scores of 0
Description: Clinical remission was defined as both rectal bleeding and stool frequency sub-scores of 0. Rectal bleeding was assessed on a scale from 0-3, where 0: no blood seen, 1: streaks of blood with stool less than half time, 2: obvious blood or streaks of blood with stool most of the time, and 3: blood alone passes. Stool frequency was assessed on a scale from 0-3, where 0: normal number of stools for this participant, 1: 1 to 2 stools more than normal, 2: 3 to 4 stools more than normal, and 3: 5 or more stools more than normal. Higher scores indicated more severe disease.
Time Frame: At Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/ Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants
  At Week 4 | 28 | 25 | 25 | 24
  At Week 8 | 22 | 25 | 29 | 31
  At Week 12 | 18 | 26 | 22 | 30
  At Week 16 | 16 | 32 | 17 | 35
  At Week 20 | 20 | 25 | 16 | 31
  At Week 24 | 12 | 31 | 12 | 31
  At Week 28 | 13 | 31 | 19 | 32
  At Week 32 | 17 | 35 | 13 | 30
  At Week 36 | 13 | 37 | 13 | 32
  At Week 40 | 15 | 34 | 12 | 25
  At Week 44 | 11 | 27 | 12 | 33
  At Week 48 | 13 | 32 | 16 | 27
  At Week 52 | 9 | 33 | 10 | 30

11. Secondary Outcome: Number of Participants With Sustained Endoscopic Remission at Week 52
Description: Sustained endoscopic remission was defined as in endoscopic remission at Week 52 visit among participants who were in endoscopic remission at the time of baseline. Endoscopic remission was defined as a centrally read endoscopic sub-score of 0 or 1 (modified, excludes friability). The centrally read endoscopic sub-score range from 0 to 3, where 0=normal or inactive disease; 3=severe disease.
Time Frame: At Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- ONTA 25mg/Placebo: PParticipants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 mg of ontamalimab were randomized to receive placebo (matched to ontamalimab) subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82
Participants | 4 | 27 | 8 | 29

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs with start dates at the time of or following the first exposure to investigational product. Number of participants with TEAEs were reported.
Time Frame: From start of study drug administration up to follow-up (Week 64)
Population: The safety set consisted of all participants who had received at least 1 dose of IP in this study, regardless of treatment received during the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]).
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg | Placebo/Placebo | Placebo/ONTA 25mg | Placebo/ONTA 75mg
Number analyzed (Participants) | 73 | 71 | 86 | 82 | 11 | 22 | 21
Participants | 46 | 41 | 54 | 51 | 8 | 11 | 12

13. Secondary Outcome: Number of Participants Who Developed Positive Antidrug Antibodies to Ontamalimab
Description: Antibody testing was conducted using an electro chemiluminescent signal method. Serum samples was analyzed for presence of antidrug antibodies to ontamalimab. Number of participants who developed positive results for ontamalimab were reported.
Time Frame: At Week 12, 24, 36 and 52
Population: The safety set consisted of all participants who had received at least 1 dose of IP in this study, regardless of treatment received during the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]). Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure and "number analyzed" refer to the participants evaluable at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | ONTA 25mg/Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg | Placebo/Placebo | Placebo/ONTA 25mg | Placebo/ONTA 75mg
Number analyzed (Participants) | 72 | 70 | 81 | 73 | 11 | 22 | 21
Participants
  At Week 12: number analyzed (Participants) | 72 | 70 | 81 | 73 | 11 | 20 | 21
  At Week 12 | 7 | 6 | 8 | 4 | 2 | 0 | 4
  At Week 24: number analyzed (Participants) | 50 | 61 | 63 | 71 | 8 | 22 | 17
  At Week 24 | 6 | 5 | 5 | 4 | 1 | 0 | 1
  At Week 36: number analyzed (Participants) | 34 | 54 | 49 | 67 | 8 | 22 | 15
  At Week 36 | 5 | 3 | 2 | 4 | 2 | 1 | 2
  At Week 52: number analyzed (Participants) | 25 | 53 | 31 | 55 | 7 | 15 | 16
  At Week 52 | 1 | 2 | 6 | 4 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 64
Groups:
- ONTA 25mg/ Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with 25 milligram (mg) of ontamalimab were randomized to receive placebo matched to ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in every 4 weeks (Q4W) up to Week 52.
- Placebo/Placebo: Participants who achieved a clinical response in one of the induction studies (SHP647-301 [NCT03259334] and SHP647-302 [NCT03259308]) with placebo were randomized to receive placebo matched to ontamalimab subcutaneously as maintenance treatment using a prefilled syringe once in Q4W up to Week 52.
Arm/Group | ONTA 25mg/ Placebo | ONTA 25mg/ONTA 25mg | ONTA 75mg/Placebo | ONTA 75mg/ONTA 75mg | Placebo/Placebo | Placebo/ONTA 25mg | Placebo/ONTA 75mg
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/71 | 1/86 | 0/82 | 1/11 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 6/73 | 9/71 | 9/86 | 2/82 | 1/11 | 0/22 | 2/21
Other Adverse Events (participants affected / at risk) | 41/73 | 27/71 | 52/86 | 30/82 | 8/11 | 11/22 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ONTA 25mg/ Placebo (N=73) | ONTA 25mg/ONTA 25mg (N=71) | ONTA 75mg/Placebo (N=86) | ONTA 75mg/ONTA 75mg (N=82) | Placebo/Placebo (N=11) | Placebo/ONTA 25mg (N=22) | Placebo/ONTA 75mg (N=21)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder metaplasia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ONTA 25mg/ Placebo (N=73) | ONTA 25mg/ONTA 25mg (N=71) | ONTA 75mg/Placebo (N=86) | ONTA 75mg/ONTA 75mg (N=82) | Placebo/Placebo (N=11) | Placebo/ONTA 25mg (N=22) | Placebo/ONTA 75mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 17 (17) | 3 (3) | 29 (34) | 6 (7) | 4 (4) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (4) | 3 (3) | 6 (7) | 2 (2) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 3 (5) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (4) | 0 (0) | 3 (3) | 1 (1) | 3 (7) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03290781/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03290781/SAP_001.pdf